CLINICAL TRIAL: NCT07298915
Title: The Effect of Exercise and Tirzepatide on Weight and Health Outcomes (EXER-MED)
Acronym: EXER-MED
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Damon Swift, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 302929
Record Dates: First submitted 2025-12-19; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight
Keywords: Obesity; Overweight; Exercise; aerobic; resistance training; GLP-1; Weight loss
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Weight Loss | interventions — Tirzepatide; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Exercise (Experimental): Participants will perform aerobic and resistance exercise while taking monthly tirzepatide for 16 weeks
  Interventions: Drug: Tirzepatide; Behavioral: Exercise
- Standard Care (Active Comparator): Participants will take monthly Tirzepatide under the care of their primary care provider for 16 weeks
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Participants will take tirzepatide under the care of their primary care provider for 16 weeks
Behavioral: Exercise — Participants will perform a combination of aerobic and resistance training for 16 weeks
  Arms: Exercise

SUMMARY:
This is clinical trials is to evaluate the effect of exercise with weight loss medication compared to weight loss alone. The study will enroll 24 adults from 30-65 years old with overweight or obesity.

The main questions it will answer includes:

* Does exercise combined with weight loss medication reduce body weight and body fat more than weight loss medication alone
* Does exercise combined with weight loss medication improve other risk factors more such as the sugar in the blood, cholesterol, fitness, and quality of life

Participants will:

* Take a weight loss medication (tirzepatide) monthly under the supervision of their primary care physician
* (Exercise group only) Will perform exercise ~3 times a week at the University of Virginia). Walking on a treadmill and resistance training
* Visit the study site at the beginning of the study and after the study to evaluate weight, body fat, and other health measures

DETAILED DESCRIPTION:
The new type class of weight loss medications called GLP-1 medications have been shown to cause weight loss and improve risk factors for heart disease and diabetes. One thing that is currently unknown is whether exercise augments the impact of weight loss in people taking GLP-1 medication. The EXER-MED study is a pilot study evaluating the effect of 16 weeks of exercise training with GLP-1 medication compared to taking the medication alone. We will evaluate the impact of the study groups on weight, body composition (percent fat, percent lean mass), blood pressure, arterial stiffness, blood work (cholesterol, blood pressure, glucose, insulin) and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 30-65 years of age, postmenopausal women included
* 27-29.9 with an additional CVD risk factor or 30-40 kg/m2
* For overweight adults only: additional cardiometabolic risk factor (diagnosed dyslipidemia, hypertension)
* Willingness and adequate health to go on weight loss medication
* The capability and willingness to provide written informed consent
* Approval of their primary care provider to go on weight loss medication

Exclusion Criteria:

* Including but not limited to serious arrhythmias
* Cardiomyopathy
* Congestive heart failure
* Stroke or transient ischemic attacks
* Peripheral vascular disease
* Previous history of myocardial infarction or stroke
* Previous diagnosis or taking medication for type 1 or 2 diabetes, fasting glucose >125 mg/dL or HbA1C ≥6.5%
* Systolic blood pressure >160 mmHg and diastolic blood pressure >100 mmHg.
* Hospitalization for mental illness within the past 5 years or currently undergoing treatment for severe mental illness
* Conditions that can be aggravated or are contraindicated by exercise training
* Plans to be out of town more than 3 weeks in the next 4 months.
* Currently pregnant or plans to become pregnant
* Currently in a diet or exercise program
* Non-compliance during screening or extreme difficulty in obtaining baseline blood samples
* Enrolled in a different exercise program
* Previous weight loss surgery
* Use of weight loss medication within the last year
* hypo/hyper thyroid (medicated or unmedicated)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Weight | Baseline and 16 Weeks
  Measurement will be taken 3 times and measured in kg. A positive value indicates an increase in weight and a negative value indicates a reduction in weight

SECONDARY OUTCOMES:
Physical activity level | Baseline and 16 weeks
  Physical activity will measured via accelerometry (total steps and light, moderate, vigorous physical activity) and steps for 7 consecutive days
Changes in Blood Lipids Concentrations | Baseline to 16 weeks
  A fasting blood sample will be used to measure low density lipoprotein, high density lipoprotein, total cholesterol, and triglycerides will be measured. It will be quantified as the specific amount of the lipoprotein within the blood in mg/dL for all lipid variables. Participants will be fasted at least 12 hours prior to the blood draw. Change will be quantified as the week 16 value subtracted from the baseline value. A positive value indicates an increase in the blood lipid variable and a negative value is associated with a reduction in the variable.
Resting Metabolic Rate | Baseline and 16 Weeks
  Resting metabolic rate (RMR) will be measured in a quiet, temperature-controlled room using indirect calorimetry with a clear ventilated canopy and dilution pump. An increase represents a positive change and a decrease represents a negative change
Change in Fasting Glucose Level | Baseline to 16 Weeks
  Change in fasting glucose level. Fasting glucose level refers to the concentration of glucose within the blood (mg/dL). The change in fasting glucose level is quantified by subtracting the week 16 value from the baseline value. Thus, a positive value indicates an increase in glucose level and a negative value indicates a decrease in glucose.
Change in Fasting Insulin Level | Baseline to 16 Weeks
  Fasting insulin represents the concentration of insulin in the blood. A positive value represents an increase in insulin concentration and a negative value represents a decrease in insulin concentration.
Change in Augmentation Index | Baseline to 16 Weeks
  Central Arterial stiffness will be measured using a SphygmoCor XCEL (Itasca, IL). Participants will refrain from large meals and caffeine for at least 2 hours and alcohol, vigorous exercise and vasoactive medication for at least 12 hours. Testing will occur in a quiet temperature controlled room in the seated position after a 5 minute rest. Augmentation index represent central arterial stiffness and will be quantified via augmentation index (%). The augmentation index (AIx) is a measure of systemic arterial stiffness, and is defined as the ratio of augmentation (Δ P) to central pulse pressure and expressed as percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. A lower value indicates better stiffness
Changes in Blood Pressure (mmHg) | Baseline to 16 weeks
  Brachial and aortic blood pressure will be measured using a sphygmocor XCEL. Blood pressure is quantified in mmHg and will be taken in the seated position after a 5 minute rest. Change in blood pressure is quantified by subtracting the week 10 value from the baseline value. Thus, a positive number is associated with an increase in blood pressure across the time point and a decrease indicates a decrease in blood pressure
Change in hemoglobin A1C | Baseline and Week 16
  Hemoglobin A1C (%) will be measured at baseline and 16 weeks. Change in hemoglobin A1C will be determined by subtracting the week 16 value from baseline. A positive change indicates and increase in hemoglobin A1C and a negative value indicates a decrease in hemoglobin A1C.
Change in Waist Circumference | Baseline to Week 16
  Waist circumference will be measured at the natural waist (midway between the inferior border of the rib cage and the superior aspect of the iliac crest) with a gulick tape measure. Both landmarks (the inferior border of the ribcage and the superior aspect of the iliac crest) will be marked and the distance will be measured to determine the appropriate measurement site. Staff will confirm that: 1) the measurement tape remains horizontal; 2) the tape touches the entire circumference of the participant; 3) abdominal tissue is not compressed; 3) the tape measure is not within abdominal folds; 4) the measurement is taken at the end of normal respiration. The measurement will be repeated an additional time, and the reported value will be the average of these measurements. Both measurements must be within 0.5 cm to be considered acceptable for data purposes. The change in waist circumference will be quantified as the the week 16 value subtracted from the baseline value
Change in Body Composition (Fat mass or Lean Mass) | Baseline to Week 16
  Dual-energy X-ray absorptiometry will be used to measure changes in fat mass and lean mass. Body fat will be quantified as the percent of fat relative to the total body composition. Lean mass will be quantified as the percent of lean tissue relative to the total body composition. Change in these variables will be quantified as by subtracting the week 16 value from the baseline value. Thus, a change in positive direction is associated with an increase in body fat or lean mass and a negative value represent a decrease.
Change in Cardiorespiratory Fitness | Baseline and 16 Weeks
  Fitness will be measured using a modified Balke protocol on a treadmill. Participants will walk at an initial speed of 2.0 mph with 0% grade for the first 3 minutes after which the treadmill speed will increase to 3.0 mph for the next 3 minutes. The treadmill grade will be increased by 2.5% every 3 minutes until volitional exhaustion. Fitness will be quantified in absolute terms (VO2) L/min, relative (VO2 mL/kg/min) and Estimated METs. Change in fitness will be quantified by subtracting the week 16 value from the baseline value. A positive value will indicate and increase in fitness. A negative value will indicate a reduction in fitness.
Change in dietary quality | Baseline to Week 16
  Dietary quality is measured with the ASA 24-hour dietary recall (ASA 24) . The ASA 24 is web-based tool that allows individuals to self-report all foods and beverages consumed in the previous 24 hours (i.e., the data collection method). This allows us to track diet quality changes over time. Change in dietary outcomes will be quantified by subtracting week 16 values from baseline. A positive value will represent an increase in a variable. A negative value will represent a reduction in a variable.
Quality of Life (IWQL-Lite) | Baseline to Week 16
  Measured by the questionnaire Impact of Weight on Quality of Life-Lite (IWQL-Lite) at baseline and Week 16. Scores range from 0 to 100, with 100 representing the best quality of life. Change in quality of life will be expressed by subtracting Week 16 from baseline level. An increase in quality of life will be represented by a positive value. A negative value represents a reduction in quality of life.
Change in isokinetic dynamometry | Baseline and Week 16
  Isokinetic knee flexor and extensor muscles strength and endurance will be evaluated with the isokinetic dynamometer. Change in strength and endurance outcomes will be quantified by subtracting the the Week 16 value from the baseline value. A positive value will indicate an increase in strength or endurance. A negative value will indicate a reduction in strength or endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Damon L Swift, Ph.D, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No